CLINICAL TRIAL: NCT01746069
Title: Evaluation of a Reinforcement Program Using Text Messages Through Mobile Phone in Smoking Cessation Programs in Primary Care
Brief Title: Effectiveness of Messages to Mobile Phone in Smoke Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Basque Health Service (Other Government)
Responsible Party: Principal Investigator, Raquel Cobos Campos, pharmaceutical, Basque Health Service
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TAB-01
Record Dates: First submitted 2012-12-07; First posted 2012-12-10 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: Smoking
Keywords: smoking; smoke cessation; sms; quit smoke
MeSH Terms: conditions — Smoking; Smoking Cessation; Smith-Magenis Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- health advice (Placebo Comparator): clinical practice routine
  Interventions: Behavioral: health advice
- Quit smoking combined cessation programme (Experimental): Health advice and support sms messages to patient's mobile phone + clinical routine practice
  Interventions: Behavioral: Quit smoking combined cessation programme

INTERVENTIONS:
Behavioral: Quit smoking combined cessation programme — Support sms messages to patient's mobile phone and health advice
  Arms: Quit smoking combined cessation programme
Behavioral: health advice — routine clinical practice
  Arms: health advice

SUMMARY:
Smoking remains a major risk factor for chronic diseases and is a real problem for health systems. The use of emerging technologies, such as mobile phone , may have a important role in smoking cessation programs through sending reinforcement messages when patients quits smoking.

Main objective: To evaluate the effectiveness of a combined 6 months smoking cessation program including health advice provided by a doctor and sending support messages to mobile phone of patients.

Methods: Study design: Randomized single blind clinical trial. Study population: Patients over 18 who are willing to start a smoking cessation program, who have mobile phone, who are able to receive and send messages, and who have a score greater than 5 or equal to 5 on the Richmond scale.

Sample size: 160 patients per arm to detect a difference in the percentage of smoking cessation than 10% (14.9% vs. 4.9%) between the two groups. Intervention: Experimental group: Health advice and support messages to mobile phone patients.

Control group: Health advice. Assessment of the primary endpoint: At 6 months (positive/negative coximetry test).

Statistical analysis: The analysis of the primary endpoint (positive / negative coximetry test) will be performed using logistic regression.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years.
* Current smoker (25): Current smoker is defined as the person who at the time of the study beginning declares that smoked daily or occasionally.
* Possessing mobile phone.
* Able to receive and send messages through mobile phone.
* Score greater than 5 or equal to 5 on the Richmond scale

Exclusion criteria:

* People with a history of mental and behavioral disorders.
* Patients with a diagnosis of depression using the depression subscale of Goldberg (two or more positive responses).
* Patients who with pharmacological therapy for smoking cessation or who require it throughout the study.
* Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2013-03; Primary Completion 2015-03 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Coximetry test (positive/negative) | at 6 months

SECONDARY OUTCOMES:
Continuous abstinence at 6 months: Yes / No | At 6 months
  Continuous Abstinence is defined as smoking more than 5 cigarettes since the beginning of the follow-up period self-reported by the patient.
Abstinence point during the first 7 days self-reported by the patient: Yes / No. | at first week
  Abstinence is defined as not smoking anything punctual during the last seven days.
-Prevalence abstinence at the 4th week self-reported by the patient: Yes / No. | At 4th week
-Prevalence abstinence at 12th week self-reported by the patient: Yes / No. | At 12th week
-Outcome of coxymetry test at 12 months of start: Positive / Negative. | at 12 months
  Only in patients with a negative result in the 6 months test
Number of messages requested by the patient anxiety. | at 12 months
slip: Yes / No. | at 12 months
  Treated as the first use (consumption point) after a period of abstinence
- Relapse: Yes / No. | At 12 months
  Relapse is defined to return dependent behavior that had tried to change, recovering or not the baseline levels before treatment.
Number of messages relapse-slip timely requested by the patient. | At 12 months

OTHER OUTCOMES:
other variables | at baseline
  Sex (male / female), age (years), number of cigarettes per day before starting program, age of start smoking (years), smoke related pathology (Yes/No), score on the anxiety scale Goldberg, previous attempts to quit smoking (Yes / No if yes, specify number of attempts and reasons for relapse), ), smoking dependence fagerström test score), type of smoker (occasional / daily).

CONTACTS AND LOCATIONS:
Locations (1):
- Health centre Lakuabizkarra, Vitoria-Gasteiz, Alava, Spain